CLINICAL TRIAL: NCT06664242
Title: Effects of TENS Application in Patients Admitted to the ICU After Cardiac Surgery: a Randomized Double-blind Clinical Trial
Brief Title: Effects of TENS in Patients Admitted to the ICU After Cardiac Surgery
Acronym: ETENSCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Max de Araujo Melo, Principal Investigator, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 76710723.0.0000.5201; 76710723.0.0000.5201 (Other: Plataforma Brasil)
Record Dates: First submitted 2024-08-30; First posted 2024-10-29 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Surgery; Transcutaneous Electric Nerve Stimulation
Keywords: tens; transcutaneous electrical nerve stimulation; heart surgery; cardiac surgical procesures; thoracic surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (Placebo Comparator): This group will not actually receive a treatment current, being subjected only to the device connected without current.
  Interventions: Device: Placebo
- TENS convencional group (Experimental): In this group, patients will undergo the hospital's usual analgesia and physiotherapy routine, plus TENS with a frequency of 140 Hz and a pulse width of 50 µs.
  Interventions: Device: Conventional TENS
- TENS low frequence group (Experimental): Patients in this group will undergo the hospital's usual analgesia and physiotherapy routine, plus conventional TENS with a low frequency of 5 Hz and a pulse width of 250 µs
  Interventions: Device: TENS low frequence group

INTERVENTIONS:
Device: Placebo — these patients will be subjected to the same usual routine of pharmacological analgesia, consisting of the administration of 1g of dipyrone at the discretion, with escalation to tramal (dose) and physiotherapy in the hospital ICU, in addition to an application of TENS, with the device turned on, with programming on channels that are not connected to the patients, so as to generate visual and auditory feedback.
  Arms: Control Group
Device: TENS low frequence group — Patients in this group will undergo the hospital usual analgesia and physiotherapy routine, in addition to conventional TENS with a low frequency of 5 Hz and a pulse width of 250 µs.
  Arms: TENS low frequence group
Device: Conventional TENS — In this group, patients will undergo the usual routine of analgesia and hospital physiotherapy, in addition to TENS with a frequency of 140 Hz, pulse width of 50 µs.
  Arms: TENS convencional group

SUMMARY:
Cardiac Surgery (CH) aims to increase survival and improve quality of life in eligible cardiac patients. However, as with any invasive intervention, pain is one of the main complaints of patients in the post-surgical period. This research is justified by the evaluation of the potential impact of the use of TENS as an alternative for analgesia in reducing the length of hospital stay and directly in the effective cost of patients undergoing cardiac surgeries, in reducing morbidity and mortality, as well as in the quality of life and early return to their daily activities, in addition to reducing the use of drugs and potentially their side effects. The objective of this study is to evaluate the effect of TENS for analgesia in hospitalized patients undergoing cardiac surgery, investigating its efficacy, safety and impact on postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes
* over 18 years of age,
* undergoing elective cardiac surgery,
* who have a sternotomy access route,
* with or without the use of pleural or mediastinal drains,
* after the first postoperative day will be selected.

Exclusion Criteria:

* with unstable angina,
* patients with arrhythmias,
* whether symptomatic or asymptomatic,
* with changes in the level of consciousness and cognition that may interfere with the assessment,
* use of metal implants,
* pacemakers and implantable cardioverter (ICD),
* those who presented postoperative complications such as infection in the sternotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
respiratory muscle strength | through study completion, an average of 1 year
  measured in centimeters of water
cough peak flow | through study completion, an average of 1 year
  measured in liters per minute
slow vital capacity | through study completion, an average of 1 year
  measured in milliliters per kilo

SECONDARY OUTCOMES:
painful sensation | through study completion, an average of 1 year
  Zero is equivalent to no pain and 10 indicates the worst possible pain.
length of stay | through study completion, an average of 1 year
  measured in days
cardiac variability | through study completion, an average of 1 year
  measured in beats per minute

CONTACTS AND LOCATIONS:
Locations (1):
- UFPE, Recife, Pernambuco, Brazil